CLINICAL TRIAL: NCT04044144
Title: Prospective Tolerability Assessment of a Probiotic Dietary Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Collaborators: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-015
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Dietary Supplement (Experimental): Subjects will be asked to take 1 capsule per day of the dietary supplement for a period of 10 days
  Interventions: Dietary Supplement: Probiotic Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Probiotic Dietary Supplement — Dietary supplement containing a combination of 8 probiotic strains

SUMMARY:
The dietary supplement being investigated is a formula containing a combination of eight probiotic strains. The combination formula was developed to support general gastrointestinal and immune health. Each of the strains in the formula have previously been studied in human subjects, including several clinical populations. However, the present eight strain combination formula has not previously been evaluated in human subjects. This prospective study will evaluate the tolerability of the eight strain formula in healthy adults.

DETAILED DESCRIPTION:
Background & Significance:

The dietary supplement being investigated is a formula containing a combination of eight probiotic strains. The combination formula was developed to support general gastrointestinal and immune health. Each of the strains in the formula have previously been studied in human subjects, including several clinical populations. However, the present eight strain combination formula has not previously been evaluated in human subjects.

Research Design & Methods:

This prospective study will evaluate the tolerability of the eight strain formula in healthy adults over a 10-day period. The primary aim of the study is to assess tolerability as determined by the frequency of study participants who withdraw from the study due to adverse events.

ELIGIBILITY:
Inclusion Criteria:

- Age 21-75 years

Exclusion Criteria:

* Currently taking a probiotic, prebiotic, or fiber supplement (or they were taken within 10 days prior to screening)
* Currently taking antibiotic, antiparasitic, or antifungal medications orally or intravenously (or they were taken within 28 days prior to screening)
* Currently taking any supplements or medications impacting gastrointestinal motility
* Active gastrointestinal infection
* Current or previous history of chronic bowel disease
* Current or previous history of liver disease
* Current or previous history of chronic kidney disease
* History of gastrointestinal surgery
* A major medical or surgical event requiring hospitalization within 3 months prior to screening
* Current or previous history of cardiovascular disease
* Current or previous history of pre-Diabetes, diabetes mellitus, or hypoglycemia
* Known infection with human immunodeficiency virus, tuberculosis, hepatitis B or hepatitis C
* Genitourinary bacterial infections within 28 days prior to screening
* Current or previous history of seizure disorder
* Current or previous history of psychiatric illness
* History of alcoholism
* Cancer within the last 5 years
* Smoking or use of nicotine containing products within 28 days prior to screening
* Use of drugs of abuse and recreational drugs/substances within 12 months prior to screening
* Known intolerance or allergy to ingredients in the study supplement
* Women who are lactating, pregnant or planning pregnancy within the next two months
* Currently participating in another interventional research study or participated in another interventional study within 28 days prior to screening

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Frequency of participants who withdraw from the study due to adverse events during the supplementation period | 0-10 days
  Tolerability of oral intake of the probiotic supplement will primarily be evaluated by determining the frequency of participants who withdraw from the study due to adverse events during the supplementation period

SECONDARY OUTCOMES:
White blood cell count | 0-10 days
  Frequency of adverse change before and after the supplementation period
Red blood cell count | 0-10 days
  Frequency of adverse change before and after the supplementation period
Hemoglobin | 0-10 days
  Frequency of adverse change before and after the supplementation period
Hematocrit | 0-10 days
  Frequency of adverse change before and after the supplementation period
Mean corpuscular volume | 0-10 days
  Frequency of adverse change before and after the supplementation period
Mean corpuscular hemoglobin | 0-10 days
  Frequency of adverse change before and after the supplementation period
Mean corpuscular hemoglobin conc. | 0-10 days
  Frequency of adverse change before and after the supplementation period
Red cell distribution width | 0-10 days
  Frequency of adverse change before and after the supplementation period
Platelet count | 0-10 days
  Frequency of adverse change before and after the supplementation period
Mean platelet volume | 0-10 days
  Frequency of adverse change before and after the supplementation period
Absolute Neutrophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Absolute Lymphocytes | 0-10 days
  Frequency of adverse change before and after the supplementation period
Absolute Monocytes | 0-10 days
  Frequency of adverse change before and after the supplementation period
Absolute Eosinophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Absolute Basophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Neutrophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Lymphocytes | 0-10 days
  Frequency of adverse change before and after the supplementation period
Monocytes | 0-10 days
  Frequency of adverse change before and after the supplementation period
Eosinophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Basophils | 0-10 days
  Frequency of adverse change before and after the supplementation period
Albumin | 0-10 days
  Frequency of adverse change before and after the supplementation period
Globulin | 0-10 days
  Frequency of adverse change before and after the supplementation period
Albumin/Globulin Ratio | 0-10 days
  Frequency of adverse change before and after the supplementation period
Alkaline Phosphatase | 0-10 days
  Frequency of adverse change before and after the supplementation period
Alanine Transaminase | 0-10 days
  Frequency of adverse change before and after the supplementation period
Aspartate Aminotransferase | 0-10 days
  Frequency of adverse change before and after the supplementation period
Blood urea nitrogen (BUN) | 0-10 days
  Frequency of adverse change before and after the supplementation period
Creatinine | 0-10 days
  Frequency of adverse change before and after the supplementation period
BUN/Creatinine ratio | 0-10 days
  Frequency of adverse change before and after the supplementation period
Calcium | 0-10 days
  Frequency of adverse change before and after the supplementation period
Carbon Dioxide | 0-10 days
  Frequency of adverse change before and after the supplementation period
Chloride | 0-10 days
  Frequency of adverse change before and after the supplementation period
Estimated Glomerular Filtration Rate | 0-10 days
  Frequency of adverse change before and after the supplementation period
Potassium | 0-10 days
  Frequency of adverse change before and after the supplementation period
Sodium | 0-10 days
  Frequency of adverse change before and after the supplementation period
Bilirubin | 0-10 days
  Frequency of adverse change before and after the supplementation period
Total Protein | 0-10 days
  Frequency of adverse change before and after the supplementation period

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Patno, PhD, Principal Investigator — Metagenics, Inc.
Locations (1):
- Personalized Lifestyle Medicine Center, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ryan JJ, Patno NM. Short-Term Tolerability, Safety, and Gut Microbial Composition Responses to a Multi-Strain Probiotic Supplement: An Open-Label Study in Healthy Adults. Integr Med (Encinitas). 2021 Feb;20(1):24-34. PMID 34393673
- See also: Full Text — http://imjournal.com/abstracts/Ryan-Short-Term-Tolerability-Safety-and-Gut-Microbial-Composition-Responses.html